CLINICAL TRIAL: NCT07407946
Title: Blended (mHealth) Trauma-Focused Cognitive Behavioral Therapy With Compassion for Adolescents With Post-Traumatic Stress Disorder: Protocol for a Pilot Randomized Controlled Trial in Northern Sweden
Brief Title: Blended Trauma-Focused Cognitive Behavioral Therapy With Compassion
Acronym: b-TF-CBT-C
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government); Region Norrbotten (Unknown); Forte (Industry); Visare Norr (Unknown); Stiftelsen Kempe-Carlgrenska Fonden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EtikDnr2024-07057-01MixadTFKBT
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Post-traumatic Stress Disorder (PTSD)
Keywords: post-traumatic stress disorder (ptsd); Adolescent; Trauma-Focused Cognitive Behavioral Therapy (TF-CBT); Blended psychotherapy; Digital mental health; mHealth intervention; Compassion-focused therapy; Self-compassion; Emotion regulation; Shame and self-criticism; Caregiver involvement; Child and adolescent psychiatry; Rural mental health; Telehealth; Pilot randomized controlled trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group, pilot randomized controlled design. Eligible adolescents are randomized in a 1:1 ratio to either the experimental blended intervention (bTF-CBT-C) or standard TF-CBT delivered in routine care. Randomization is stratified by geographic region and uses permuted blocks to ensure balance between groups. Participants remain in their assigned group throughout the study, and outcomes are assessed concurrently across groups at predefined time points.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of psychological treatment, participants and care providers cannot be blinded to group assignment. Outcome assessors are blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended TF-CBT with Compassion (bTF-CBT-C) (Experimental): Participants assigned to this arm receive blended trauma-focused cognitive behavioral therapy with integrated compassion-focused strategies (bTF-CBT-C), delivered in a structured sequence combining therapist-led sessions and self-paced app-based modules. The intervention includes an initial clinic-based introduction with safety planning (C0), app-supported psychoeducation and compassion-based stabilization modules targeting emotion regulation and compassionate coping (C1-C5), therapist-led trauma narrative and cognitive processing delivered via videoconferencing and selected in-person sessions (C6), followed by in vivo mastery, conjoint caregiver-adolescent work, and future-oriented relapse prevention and recovery planning (C7-C9).
  Caregiver involvement follows TF-CBT principles and compassion-focused strategies and is integrated throughout treatment. Caregivers participate in the initial session and safety planning, complete parallel app-based modules during the stabilization phase.
  Interventions: Behavioral: Blended Trauma-Focused Cognitive Behavioral Therapy with Compassion (bTF-CBT-C)
- Standard Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) (Active Comparator): Participants assigned to this arm receive standard trauma-focused cognitive behavioral therapy (TF-CBT) delivered face-to-face and through videoconference in routine child and adolescent psychiatric care. Treatment follows the TF-CBT PRACTICE components, including psychoeducation, emotion regulation skills, cognitive coping, trauma narrative and processing, in vivo exposure, conjoint caregiver-adolescent sessions, and safety planning, with caregiver involvement according to the TF-CBT manual.
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT)

INTERVENTIONS:
Behavioral: Blended Trauma-Focused Cognitive Behavioral Therapy with Compassion (bTF-CBT-C) — Blended trauma-focused cognitive behavioral therapy with integrated compassion-focused strategies, combining therapist-led videoconferencing and selected in-person sessions with self-paced app-based modules. The intervention includes an initial introduction and safety planning, a stabilization phase with digital psychoeducation and compassion-based emotion regulation skills, therapist-led trauma narrative and cognitive processing, and a recovery phase focusing on in vivo mastery, caregiver-adolescent conjoint work, and relapse prevention. Caregivers participate throughout treatment, including parallel app-based modules during stabilization and selected therapist-led sessions.
  Other Names: bTF-CBT-C; Blended TF-CBT with Compassion
  Arms: Blended TF-CBT with Compassion (bTF-CBT-C)
Behavioral: Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) — Standard trauma-focused cognitive behavioral therapy delivered face-to-face in routine child and adolescent psychiatric care. Treatment follows the TF-CBT PRACTICE components, including psychoeducation, affect regulation, cognitive coping, trauma narrative and processing, in vivo exposure, conjoint caregiver-adolescent sessions, and safety planning, with caregiver involvement according to the TF-CBT manual.
  Other Names: TF-CBT
  Arms: Standard Trauma-Focused Cognitive Behavioral Therapy (TF-CBT)

SUMMARY:
Brief Summary

The goal of this clinical trial is to evaluate the feasibility and acceptability of a blended (mHealth) Trauma-Focused Cognitive Behavioral Therapy with Compassion (bTF-CBT-C) for adolescents with post-traumatic stress disorder (PTSD) in routine child and adolescent psychiatric services in northern Sweden. The main questions it aims to answer are:

* Is bTF-CBT-C feasible to deliver in routine care, as indicated by recruitment, retention, adherence to sessions and app modules, data completeness, and adverse events?
* Is bTF-CBT-C acceptable to adolescents, caregivers, and therapists, as indicated by satisfaction, therapeutic alliance, digital treatment evaluation, and qualitative interviews? Researchers will compare bTF-CBT-C to standard TF-CBT to explore whether the blended format shows similar or potentially improved patterns in clinical outcomes (e.g., PTSD symptoms, emotion regulation, and self-compassion) and to estimate variability needed to plan a future non-inferiority trial.

Participants will:

* Complete eligibility screening and baseline assessments, including a diagnostic interview for PTSD.
* Be randomized to either bTF-CBT-C or standard TF-CBT.
* Receive trauma-focused treatment over time, with caregiver involvement in both groups.
* In the bTF-CBT-C group, use a secure mobile app for stabilization modules and exercises, together with therapist-led video sessions and selected in-person meetings.
* Complete assessments at baseline, after stabilization, post-treatment, and at 6-month follow-up, and provide feedback about their experiences (questionnaires and interviews).

DETAILED DESCRIPTION:
Detailed Description This study is a two-arm, parallel-group, pilot randomized controlled trial designed to evaluate the delivery of a blended (mHealth) Trauma-Focused Cognitive Behavioral Therapy with Compassion (bTF-CBT-C) for adolescents with post-traumatic stress disorder (PTSD) within routine child and adolescent psychiatric services in northern Sweden. The trial primarily targets feasibility and acceptability of trial procedures and intervention delivery in real-world clinical settings, and will generate preliminary estimates of variability in key clinical and mechanism-related measures to inform the design of a subsequent fully powered non-inferiority trial.

Design and setting The trial will be conducted in publicly funded child and adolescent psychiatry (CAP) clinics in Regions Västerbotten and Norrbotten, Sweden. Participants will be randomized 1:1 to bTF-CBT-C (experimental) or standard TF-CBT (control). Randomization will be generated by an independent researcher using permuted blocks (block size 4) and stratified by geographic region. Allocation concealment will be maintained using sequentially numbered sealed opaque envelopes. Due to the nature of psychological treatment, participants and therapists cannot be blinded.

Intervention rationale and structure Standard TF-CBT is the recommended first-line psychological treatment for youth PTSD, but access in rural regions is challenged by long travel distances and limited therapist availability. bTF-CBT-C has been developed to reduce structural barriers while maintaining therapeutic alliance and emotional safety, with particular attention to shame and self-criticism commonly present after interpersonal trauma. The intervention follows the TF-CBT PRACTICE framework and integrates compassion-focused strategies intended to support engagement and reduce threat-based responding during trauma-focused work.

Experimental arm: bTF-CBT-C (blended TF-CBT with compassion) bTF-CBT-C combines (1) an initial therapist-led clinic session, (2) self-paced app-based stabilization modules with between-session practice, (3) therapist-led videoconferencing sessions, and (4) selected in-person sessions when clinically indicated. The intervention is delivered across three overarching phases:

1. Stabilization (Modules C0-C5): app-based psychoeducation and skills training for adolescents and caregivers (e.g., emotion regulation strategies and compassion-based practices such as soothing rhythm breathing and compassionate imagery). The stabilization phase is supported by therapist check-ins (video) and clinic routines, and includes an individualized safety plan developed together with the adolescent and caregiver.
2. Trauma processing (Module C6): therapist-led trauma narration and cognitive processing using TF-CBT procedures, delivered primarily via secure videoconferencing and supplemented with in-person sessions as needed. Compassion-focused strategies are used to address shame and self-criticism and to support emotional safety and approach behavior during trauma-focused work.
3. Integration and recovery (Modules C7-C9): consolidation of gains, in-vivo mastery/exposure planning where relevant, conjoint caregiver-adolescent work, and future-oriented relapse prevention supported by compassionate imagery and values-consistent planning.

The digital components are delivered using the CE-marked Amnicare mobile application. Videoconferencing is delivered via GDPR-compliant platforms used in routine care (e.g., Visiba Care and Platform24). Participants use their own smartphone/tablet; technical support is available through the clinic.

Control arm: standard TF-CBT Participants allocated to the control arm receive standard TF-CBT delivered face-to-face and with videoconference in routine care by clinicians trained in TF-CBT, including the core PRACTICE components and caregiver involvement in line with the manual. Usual clinical flexibility regarding number of sessions and pacing is retained, consistent with routine care delivery.

Assessments and follow-up The trial includes assessments at baseline, after completion of the stabilization phase, post-treatment, and at 6-month follow-up. In addition, brief weekly process measures are collected during the intervention period to capture engagement, alliance, usability/experience of digital components (where applicable), and key mechanism-relevant processes (e.g., shame/guilt-related responses). Qualitative interviews with adolescents, caregivers, and therapists are conducted during and/or after treatment to capture experiences of the blended format, perceived helpfulness and burden, and recommendations for refinement.

Safety and risk management A structured safety plan is developed with each adolescent and caregiver prior to the digital stabilization phase. Risk and emotional safety are monitored weekly through brief self-report items. Any indication of increased risk triggers clinician follow-up according to routine CAP procedures. Videoconferencing sessions follow a predefined protocol for interrupted calls (immediate reconnection attempts, phone contact, and escalation to welfare checks/emergency procedures as clinically indicated). Adverse events and serious adverse events are documented in a study safety log and reviewed in supervision.

Data management and confidentiality Study data are pseudonymized and stored on secure, access-restricted servers. Data transfer from digital components uses encrypted channels and complies with GDPR and institutional requirements for sensitive personal data. Only authorized members of the research team have access to identifiable data.

Statistical approach (pilot focus) Analyses will follow intention-to-treat principles. Feasibility and acceptability indicators will be summarized descriptively (e.g., proportions, means, and confidence intervals). Exploratory models (e.g., baseline-adjusted ANCOVA and/or mixed-effects models) will be used to describe symptom trajectories and estimate variability and preliminary effect size ranges for planning the future non-inferiority trial; the study is not powered for formal effectiveness testing. Qualitative interviews will be analyzed using reflexive thematic analysis.

Progression criteria Predefined progression criteria will guide decisions about moving to a fully powered non-inferiority trial, focusing on recruitment, retention, acceptability, and data completeness thresholds consistent with pilot and feasibility trial guidance. Findings will be used to refine trial procedures, therapist training/support, and the blended intervention structure prior to scale-up.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-17 years.
* Meet DSM-5 criteria for post-traumatic stress disorder (PTSD) confirmed by diagnostic interview (MINI-KID).
* Score ≥25 on the Child and Adolescent Trauma Screen (CATS-2) at baseline.
* Receiving care within routine child and adolescent psychiatric services in participating regions.
* Have a non-offending caregiver willing and able to participate in caregiver components of treatment.
* Able to communicate in Swedish sufficiently to engage in treatment and assessments.
* Provide informed assent/consent, with caregiver consent according to age and regulations.

Exclusion Criteria:

* Acute suicidality or risk requiring inpatient care.
* Active psychotic disorder or severe dissociative symptoms that interfere with participation.
* Autism spectrum disorder, severe eating disorder, or obsessive-compulsive disorder requiring primary specialized treatment.
* Ongoing trauma exposure or unstable living conditions that would prevent safe participation.
* Cognitive impairment or medical condition that precludes participation in psychotherapy or digital components.
* Substance use disorder requiring treatment, or regular use of benzodiazepines (> once per week).
* Concurrent trauma-focused psychotherapy or recent initiation/discontinuation of psychotropic medication (within the past 6 weeks), or planned medication changes during the study period.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline (enrollment, day 1)
  Proportion of eligible adolescents who consent to participate.
Retention Rate | Baseline (day 1), poststabilization (completion after an average of 5 weeks), post-treatment (study completion up to 25 weeks) up to 6 months
  Proportion of enrolled participants completing post-stabilization, post-treatment, and 6-month follow-up assessments.
Adherence to Treatment Components | Post-stabilization (an average of 5 weeks) and post-treatment (study completion up to 25 weeks).
  Adherence will be assessed as (1) the number of therapist-led sessions attended out of the planned total, and (2) the number of app-based modules (C0-C9) completed. Higher numbers reflect higher adherence.
Adverse Events | From baseline through treatment completion (up to 25 weeks) to 6 months follow up after study completion.
  Number and type of adverse events reported during the intervention.
Acceptability and User Experience (Qualitative Interviews) | Through study completion, up to 6 month follow up.
  Semi-structured qualitative interviews will explore overall acceptability, perceived helpfulness, usability, burden, and user experience of the blended TF-CBT with compassion.

SECONDARY OUTCOMES:
Treatment Satisfaction | Post-treatment, study completion (up to 25 weeks).
  Overall treatment satisfaction will be assessed using a single-item rating scale where adolescents rate their satisfaction with the blended TF-CBT with compassion. Higher scores indicate greater satisfaction.
Therapeutic Alliance | Post-treatment, study completion (up to 25 weeks).
  Therapeutic alliance will be assessed using a brief alliance scale based on goals, tasks, and bond. Higher scores indicate stronger alliance.
Post-traumatic stress disorder symptoms | Baseline, Post-stabilization (an average of 5 weeks), Post-treatment (study completion up to 25 weeks) and Follow-up (6 months after treatment completion)
  PTSD symptoms will be assessed using the Child and Adolescent Trauma Screen (CATS-2). CATS-2 includes three subscales: (1) Traumatic Events (15 items, score range 0-15; higher scores indicate more trauma exposure), (2) Posttraumatic Stress Symptoms (20 items, score range 0-60; higher scores indicate more severe PTSD symptoms), and (3) Functional Impairment (5 items, score range 0-5; higher scores indicate greater impairment).
Post-traumatic stress disorder symptoms | Baseline, Post-stabilization (an average of 5 weeks), Post-treatment (study completion up to 25 weeks) and Follow-up (6 months after treatment completion)
  Post-traumatic stress symptoms will also be assessed using the Children's Revised Impact of Event Scale - 13 items (CRIES-13). The CRIES-13 includes 13 items rated on a 4-point scale (0 = not at all, 1 = rarely, 3 = sometimes, 5 = often), with a total score range of 0-65. The scale comprises three subscales: Intrusion, Avoidance, and Arousal. Higher scores indicate more severe post-traumatic stress reactions. A total score ≥30 is considered indicative of clinically significant PTSD risk.
Emotion regulation difficulties | Baseline, Post-stabilization (an average of 5 weeks), Post-treatment (study completion up to 25 weeks) and Follow-up (6 months after treatment completion)
  Emotion regulation will be assessed using the Difficulties in Emotion Regulation Scale - 16 item version (DERS-16). The DERS-16 contains 16 items rated on a 5-point Likert scale (1 = almost never to 5 = almost always), yielding a total score range of 16-80. Higher scores indicate greater difficulties in emotion regulation. The measure includes five subscales: Clarity, Goals, Impulse, Strategies, and Nonacceptance.
Self-compassion | Baseline, Post-stabilization (an average of 5 weeks), Post-treatment (study completion up to 25 weeks) and Follow-up (6 months after treatment completion)
  Self-compassion will be assessed using the Compassionate Engagement and Action Scales for Youth, Swedish version (CEASY-SE). The CEASY-SE is a 27-item self-report measure assessing compassion across three scales: Self-Compassion, Compassion for Others, and Compassion from Others, each consisting of Engagement and Action subcomponents. Items are rated on a Likert scale, and subscale scores are summed, with higher scores indicating greater compassion competencies.
Depression | Baseline, Post-stabilization (an average of 5 weeks), Post-treatment (study completion up to 25 weeks) and Follow-up (6 months after treatment completion)
  Depressive symptoms and suicidality will be assessed using the Montgomery-Åsberg Depression Rating Scale for Youth (MADRS-Y). The MADRS-Y is a 12-item self-report scale rated from 0 to 6 per item, yielding a total score range of 0-72. Higher scores indicate more severe depressive symptoms.
Dissociative symptoms | Baseline, Post-stabilization (an average of 5 weeks), Post-treatment (study completion up to 25 weeks) and Follow-up (6 months after treatment completion)
  Dissociative symptoms will be assessed using the Dissociation Screening Questionnaire (DSQ-12). The DSQ-12 is a 12-item self-report measure assessing psychoform and somatoform dissociation. Items are rated on a 5-point scale (0 = never to 4 = always), yielding a total score range from 0 to 48. Higher sco
Depression and anxiety | Baseline, Post-stabilization (an average of 5 weeks), Post-treatment (study completion up to 25 weeks) and Follow-up (6 months after treatment completion)
  Anxiety and depressive symptoms will be assessed using the Revised Child Anxiety and Depression Scale - 47-item version (RCADS-47). The RCADS-47 contains 47 items rated on a 4-point Likert scale (0 = never to 3 = always). It yields six subscale scores: Separation Anxiety Disorder, Social Phobia, Generalized Anxiety Disorder, Panic Disorder, Obsessive-Compulsive Disorder, and Major Depressive Disorder. A Total Anxiety score (sum of the five anxiety subscales) and a Total Internalizing score (sum of all six subscales) are also calculated. Higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Inga Dennhag, PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Clinical Science, Child- and Adolescent Psychiatry, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the sensitive nature of the data, the inclusion of minors, and ethical and legal restrictions related to confidentiality and data protection. De-identified aggregate data may be shared in publications and upon reasonable request, subject to ethical approval and applicable data protection regulations.

REFERENCES:
- [Background] Wallin, L., Svedin, C.-G., Wiberg, M., & Dennhag, I. (2026). The Compassionate Engagement and Action Scale for Youths: psychometric properties in a clinical psychiatric Swedish sample [Original Research]. Frontiers in Psychology, Volume 16 - 2025. https://doi.org/10.3389/fpsyg.2025.1653979
- [Background] Wallin, L., Lundqvist, U., Svedin, C.-G., & Dennhag, I. (2024). "Longing to be cared about and cared for" Exploring Experiences of Trauma Therapy and Views on Future Trauma Therapy (Including Digital) for Young People in Rural Northern Sweden. Children and Youth Services Review, 166, 107953. https://doi.org/https://doi.org/10.1016/j.childyouth.2024.107953
- [Background] Vestin, M., Wallin, L., Naesstrom, M., Blomqvist, I., Svedin, C. G., Beaumont, E., Jokinen, J., & Dennhag, I. (2025). Internet-based group compassion-focused therapy for Swedish young people with stress, anxiety and depression: a pilot waitlist randomized controlled trial. Frontiers in Psychology, 16(1547046), 1547046. https://doi.org/10.3389/fpsyg.2025.1547046
- [Background] Cohen, J., Mannarino, A., & Deblinger, E. (2017). Treating trauma and traumatic grief in children and adolescents. (2 ed.). The Guilford Press.
- Available data/document: Homepage at Umeå University in Sweden — https://www.umu.se/forskning/projekt/utveckling-och-behandling-av-compassionfokuserad-internetformedlad-tf-kbt-for-ungdomar-med-posttraumatisk-stress/